CLINICAL TRIAL: NCT05428644
Title: The Effect of Massage on Patients Undergoing Coronary Artery Bypass Graft Surgery
Brief Title: Effect of Reflexology Massage on Pain and Anxiety.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gizem Göktuna, Principal Investigator, Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 2021/04-24 08.02.2021
Record Dates: First submitted 2022-03-23; First posted 2022-06-23 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Pain; Anxiety
Keywords: hand reflexology; nursing care; pain management
MeSH Terms: conditions — Pain; Anxiety Disorders; Agnosia | interventions — Massage

STUDY DESIGN:
Intervention Model Description: A double-blind randomised controlled clinical trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reflexology hand massage group (Active Comparator): In addition to the standard nursing care of the hospital, individuals in the reflexology hand massage will be given a 10-minute massage for both hands, a total of 20 minutes, after the extubation procedure.
  Interventions: Behavioral: massage therapy
- placebo hand massage group (Placebo Comparator): In addition to the standard nursing care of the hospital, individuals in the placebo hand massage group will be given a 10-minute massage for both hands, a total of 20 minutes, after the extubation procedure.
  Interventions: Behavioral: massage therapy

INTERVENTIONS:
Behavioral: massage therapy — In addition to the standard nursing care of the hospital, individuals in the reflexology hand massage and placebo hand massage group will be given a 10-minute massage for both hands, a total of 20 minutes, after the extubation procedure.

SUMMARY:
Aim: The aim of this study is to examine the effects of reflexology hand massage group and placebo group on pain and anxiety in patients undergoing coronary artery bypass graft surgery.

Method: Individuals who have undergone coronary artery bypass graft surgery in accordance with the sampling inclusion criteria will be allocated to the reflexology and placebo groups by block randomization using the randomization method. After the groups are determined, the patients in the reflexology hand massage group and placebo group will be asked to fill in the Socio-Demographic Information Form, the State Anxiety Scale and the Visual Analog Scale will be taken.

In addition to the standard nursing care of the hospital, individuals in the reflexology group and placebo group will be massaged for 10 minutes, a total of 20 minutes, after the extubation procedure. Individuals in the reflexology group and placebo group will be followed up before the massage (0. minute) and after the massage at the 5th, 30th and 60th minutes, and the data will be recorded.

DETAILED DESCRIPTION:
Pain and anxiety are common postoperative problems that impair recovery and quality of life in patients undergoing coronary artery bypass graft (CABG) surgery. These problems cause changes in physiological parameters, prolonged recovery, sleep problems and a decrease in quality of life in patients. Hand reflexology, which is among the non-pharmacological methods, is an effective intervention that nurses can apply independently in the management of pain and anxiety.Therefore, this study aimed to examine the effect of reflexology on pain and anxiety.

ELIGIBILITY:
Inclusion Criteria:

* To be over 18 years of age,
* To know Turkish and to agree to participate in the research
* No previous open heart surgery
* Non-urgent planned bypass surgery
* Without any intra-aortic balloon pump or pacemaker
* Not taking inotropic drugs
* Patients who have no problem to apply massage; Those who do not have any skin lesions, burns
* Extubated
* Not taking analgesics

Exclusion Criteria:

* Mitral valve repair or replacement during CABG surgery
* Those who have any skin lesions, burns, open wounds, muscle and bone-related pathological disease, phlebitis
* Not disconnected from mechanical ventilation
* Having a risk factor for complications (e.g: ejection fraction < 35%)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
pain scores of reflexology hand massage and placebo hand massage group | Individuals in the reflexology hand massage and placebo hand massage groups will be monitored up before the massage.
  Comparison of pain scores between reflexology hand massage and placebo hand massage groups. The patients' pain score data were collected by the Visual Analog Scale. It is a 10-point scale. Higher points show a higher level of pain.
pain scores of reflexology hand massage and placebo hand massage group | Individuals in the reflexology hand massage and placebo hand massage groups will be monitored up 5th minute after the massage.
  Comparison of pain scores between reflexology hand massage and placebo hand massage groups. The patients' pain score data were collected by the Visual Analog Scale. It is a 10-point scale. Higher points show a higher level of pain.
pain scores of reflexology hand massage and placebo hand massage group | Individuals in the reflexology hand massage and placebo hand massage groups will be monitored up 30th minute after the massage.
  Comparison of pain scores between reflexology hand massage and placebo hand massage groups. The patients' pain score data were collected by the Visual Analog Scale. It is a 10-point scale. Higher points show a higher level of pain.
pain scores of reflexology hand massage and placebo hand massage group | Individuals in the reflexology hand massage and placebo hand massage groups will be monitored up 60th minute after the massage.
  Comparison of pain scores between reflexology hand massage and placebo hand massage groups. The patients' pain score data were collected by the Visual Analog Scale. It is a 10-point scale. Higher points show a higher level of pain.

SECONDARY OUTCOMES:
anxiety scores of reflexology hand massage and placebo hand massage group | Individuals in the reflexology hand massage and placebo hand massage groups will be followed up before the massage.
  Comparison of anxiety scores between reflexology hand massage and placebo hand massage groups. The patients' anxiety score data were collected by the State Anxiety Inventory. It is a 20-item scale. The scores in the inventory range from 20 to 80. Higher points show a higher level of anxiety.
anxiety scores of reflexology hand massage and placebo hand massage group | Individuals in the reflexology hand massage and placebo hand massage groups will be monitored up 60th minute after the massage.
  Comparison of anxiety scores between reflexology hand massage and placebo hand massage groups. The patients' anxiety score data were collected by the State Anxiety Inventory. It is a 20-item scale. The scores in the inventory range from 20 to 80. Higher points show a higher level of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Gülşah Gürol Arslan, PhD, Principal Investigator — Associate professor
Locations (1):
- Dokuz Eylül University, Balçova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No